CLINICAL TRIAL: NCT00815360
Title: Ranibizumab (rhuFab V2) and Scatter Laser Photocoagulation in Treatment of Patients With Clinically-significant Diabetic Macular Edema With Peripheral Retinal Nonperfusion (RaScaL)
Brief Title: Ranibizumab and Peripheral Scatter Laser in Patients With Diabetic Macular Edema and Peripheral Nonperfusion
Acronym: RaScaL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Retina Associates of Florida, P.A. (Other)
Responsible Party: Principal Investigator, Ivan J. Suner, MD, Director of Clinical Research, Retina Associates of Florida, P.A.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00002813
Record Dates: First submitted 2008-12-26; First posted 2008-12-30 (Estimated); Results first posted 2015-03-05 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2014-10

CONDITIONS: Diabetic Macular Edema
Keywords: diabetic macular edema

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment group (Experimental): 1. single intravitreal injection of ranibizumab (0.5 mg in 0.1 cc)
  2. peripheral laser to areas of retinal nonperfusion on ultra-widefield fluorescein angiography
  Interventions: Drug: intravitreal injection of ranibizumab; Procedure: peripheral laser
- Control Group (Active Comparator): 1. single intravitreal injection of triamcinolone acetonide (4.0 mg in 0.1 cc)
  2. macular laser per treatment criteria
  Interventions: Drug: intravitreal injection of triamcinolone acetonide; Procedure: macular laser

INTERVENTIONS:
Drug: intravitreal injection of ranibizumab — intravitreal injection of 0.5 mg ranibizumab
  Other Names: treatment arm
  Arms: Treatment group
Procedure: peripheral laser — ultra-widefield fluorescein angiography guided peripheral laser
  Other Names: treatment arm
  Arms: Treatment group
Drug: intravitreal injection of triamcinolone acetonide — intravitreal injection of 4.0 mg triamcinolone acetonide
  Other Names: control arm
  Arms: Control Group
Procedure: macular laser — macular laser to areas of retinal thickening or leakage
  Other Names: control arm
  Arms: Control Group

SUMMARY:
To investigate the role of ranibizumab and angiographically-directed peripheral scatter laser therapy in patients with clinically-significant diabetic macular edema (CSME) and peripheral nonperfusion. We propose a novel treatment of CSME in a subgroup of patients defined by a combination of ultrawide-field angiography (UWFA) and optical coherence tomography (OCT). Within this classification scheme, patients with CSME are subdivided by the presence of: 1) focal macular leakage, 2) vitreomacular interface traction, and/or 3) peripheral nonperfusion. The successful treatment of diabetic macular edema would be dictated by pathophysiology-directed therapy based on this classification.

The subgroup of interest for this clinical trial is characterized by diabetic macular edema, peripheral nonperfusion on UWFA, and the absence of macular traction on OCT. This group of patients has previously not been well recognized or characterized due to limitations in previous, standard angiographic evaluation of the retinal periphery.

We postulate that this subcategory represents one with a high rate of failure of accepted therapies given persistence of the basic pathophysiologic mechanism for CSME, namely ischemia-induced production of Vascular Endothelial Growth Factor (VEGF) from the retinal periphery. This also represents a population of patients with likely recurrence of CSME despite treatment with anti-VEGF therapy alone for the same reason.

DETAILED DESCRIPTION:
Diabetic retinopathy is a leading cause of moderate and severe visual loss in developed countries. It is of paramount socioeconomic impact as the prevalence of diabetes is sharply increasing, diabetic macular edema is the leading cause of vision loss in working age patients, it is a significant cause of vision loss in patients older than 65 years of age, it frequently affects patients bilaterally, and the costs of therapy are increasing.

Diabetic macular edema (DME) is the most common cause of vision loss in diabetic retinopathy. The pathophysiology of DME is complex and multifactorial. Chronic hyperglycemia, protein kinase C (PKC) formation, free radical accumulation, advanced glycation end-product (AGE) proteins, and ischemia-driven release of vascular endothelial growth factor (VEGF) are some of the better understood factors that contribute to chronic retinal arterial and capillary damage and increased permeability.

The RIDE and RISE Studies demonstrated the superiority of anti-VEGF monotherapy with ranibizumab over sham therapy, when all groups were allowed to receive macular laser therapy after month 3 based on predefined criteria. Furthermore, other studies have demonstrated VEGF inhibitors to be beneficial for DME, either as monotherapy or in combination with macular laser.

The benefit of VEGF antagonists in treating DME validates that the VEGF pathway is a key target. The need for repeated anti-VEGF injections to maintain the benefit of treatment begs the question whether persistent peripheral retinal ischemia may be driving VEGF production in at least a subset of patients with DME. Fluorescein angiographic studies of the mid- and far-periphery of diabetic patients by Shimizu in the 1980's demonstrated areas of peripheral retinal nonperfusion in diabetic patients. These findings have been reproduced and substantiated more recently utilizing a novel, commercially-available imaging system for ultrawide-field angiography (UWFA) that employs a scanning laser ophthalmoscope and an ellipsoidal mirror.

We investigated whether patients with diabetic macular edema associated with peripheral nonperfusion on UWFA would have improved visual acuity, resolution of retinal thickening on OCT, and durability of therapy using a novel strategy of a single intravitreal injection of Ranibizumab, a VEGF-A inhibitor + UWFA-guided peripheral Scatter Laser, or RaScaL. A second goal of the study was to guide DME treatment by the imaging signature of UWFA and OCT.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible if the following criteria are met:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 18 years

Patient related considerations:

• Patients with Type I or Type II diabetes

Disease related considerations:

* Study eye with clinically significant diabetic macular edema characterized by macular edema, peripheral nonperfusion, and absence of macular traction on clinical exam, UWFA, and OCT.
* Study eye with best corrected visual acuity between 20/40 (≤ 73 letters on Early Treatment of Diabetic Retinopathy Study (ETDRS) chart and 20/320 (≥ 19 letters on ETDRS chart) Other considerations
* Patient able to complete all study visits
* Female patients must be using two forms of contraception

Exclusion Criteria:

* Pregnancy (positive pregnancy test) or lactation. Premenopausal women not using adequate contraception. The following are considered effective means of contraception: surgical sterilization or use of oral contraceptives, barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel, an Intra Uterine Device, or contraceptive hormone implant or patch.
* Prior enrollment in the study
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
* Participation in another simultaneous medical investigation or trial
* Therapy with intravitreal triamcinolone, pegaptanib, ranibizumab, or bevacizumab within the previous 3 months
* Previous panretinal scatter laser photocoagulation
* Previous pars plana vitrectomy
* Visually-significant significant cataracts as primary reason for vision loss
* Uncontrolled or advanced glaucoma
* Patients on more than one anti-glaucoma agent
* Myocardial infarction or cerebrovascular accident within 6 months
* Subjects with poor glycemic control that have initiated intensive insulin treatment or plan to do so in the next 4 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-02; Primary Completion 2011-07 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivan J Suner, MD, Principal Investigator — Retina Associates of Florida
Locations (1):
- Retina Associates of Florida, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We included 30 treatment-naïve eyes of 22 patients (8 bilateral patients) aged ≥ 18 years of age, with Type 1 or 2 diabetes mellitus and visual impairment secondary to diabetic macular edema associated with peripheral nonperfusion on Ultra Widefield Fluorescein Angiography (UWFA).
Pre-assignment Details: Treatment naive patients
Groups:
- Treatment Group 1: ranibizumab and scatter laser
- Comparative Group 1: Intravitreal triamcinolone with macular laser
Period: Overall Study
Arm/Group | Treatment Group 1 | Comparative Group 1
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group 1 | Comparative Group 1 | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 11 | 21
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (7.5) | 58.3 (6.5) | 58.0 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 6 | 6 | 12
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Best Corrected Visual Acuity (BCVA), as Assessed by the Number of Letters Read Correctly on the ETDRS Eye Chart at a Starting Test Distance of 4 Meters From Baseline to Month 6.
Time Frame: 6 months
Population: We included 30 treatment-naïve eyes of 22 patients (8 bilateral patients) aged ≥ 18 years of age, with Type 1 or 2 diabetes mellitus and visual impairment secondary to diabetic macular edema associated with peripheral nonperfusion on UWFA.
Measure: Mean (95% Confidence Interval); unit: Letters of visual acuity on ETDRS chart
Units Other Than Participants: Eyes
Arm/Group | Treatment Group 1 | Comparative Group 1
Number analyzed (Participants) | 11 | 11
Number analyzed (Eyes) | 15 | 15
Letters of visual acuity on ETDRS chart | 13 [9 to 15] | 10 [7 to 13]

2. Secondary Outcome: Mean Central Foveal Thickness (CFT) on Optical Coherence Tomography (OCT) in Microns at 6 Months
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: units on a scale (microns)
Units Other Than Participants: Eyes
Arm/Group | Treatment Group 1 | Comparative Group 1
Number analyzed (Participants) | 11 | 11
Number analyzed (Eyes) | 15 | 15
units on a scale (microns) | 270 [240 to 310] | 350 [280 to 400]

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- Treatment Group 1: Intravitreal ranibizumab and peripheral laser
- Comparative Group 1: Intravitreal triamcinolone acetonide and macular laser
Arm/Group | Treatment Group 1 | Comparative Group 1
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

LIMITATIONS AND CAVEATS:
small study size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No